CLINICAL TRIAL: NCT06047613
Title: Inflammation and Blood Brain Barrier Integrity as Biomarkers of Suicidal Behavior
Acronym: IBBBiS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0103
Record Dates: First submitted 2023-07-21; First posted 2023-09-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Suicide; Depression
Keywords: suicide; depression
MeSH Terms: conditions — Suicide; Depression | interventions — Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suicide attempters (Experimental): Currently depressed patients with a suicide attempt within the 8 last days (with a maximal lifetime number of 3 previous suicide attempt including the most recent );
  Interventions: Biological: Blood samples; Other: Hetero-questionnaires and auto-questionnaires; Other: Magnetic Resonance Imaging (MRI)
- Affective controls (Active Comparator): Currently depressed patients without any lifetime history of suicide attempt
  Interventions: Biological: Blood samples; Other: Hetero-questionnaires and auto-questionnaires; Other: Magnetic Resonance Imaging (MRI)
- Healthy controls (Active Comparator): Participants with no lifetime history of psychiatric disorders
  Interventions: Biological: Blood samples; Other: Hetero-questionnaires and auto-questionnaires; Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Biological: Blood samples — Blood samples will be collected at both visit between 8:30 a.m. and 10 a.m. and fasting from midnight.
Other: Hetero-questionnaires and auto-questionnaires — Questionnaires will be administrated at both visits to assess the suicide spectrum, the depression level and some personality traits.
  Heteroquestionnaires will be administrated during a clinical interview (1h) conducted by a psychiatrist or psychologist. Autoquestionnaires (45 min) will be completed by the participant himself.
Other: Magnetic Resonance Imaging (MRI) — MRI will be processed (at both visits for patients and at inclusion visit for healthy controls) to study between groups white matter microstructure and brain functional connectivity networks

SUMMARY:
Recent studies have revealed an association between history of suicide attempt and inflammatory markers in both the cerebrospinal fluid and the plasma. Post mortem studies have shown an increase in microglial activation in the brain tissue of suicide victims. However the relationship between peripheral and central inflammation in suicide is probably mediated by complex biological processes that are yet elucidated. An increase of blood S100B levels (biomarker of neurovascular damage; PMID 14530574) has been reported in adolescents with suicidal ideation vs. controls and independently of psychiatric disorder.

The investigators hypothesize that peripheral inflammation may alter the blood brain barrier, which normally acts as a filter to ensure proper neuronal functioning, in suicidal patients.

They propose to investigate peripheral inflammation, neurovascular permeability and miRNAs in suicidal behavior pathophysiology as biomarkers of suicidal behavior in depression

DETAILED DESCRIPTION:
150 participants will be enrolled, divided into 3 groups:

* 50 Suicide attempters, i.e. currently depressed patients with a suicide attempt within the 8 last days (with a maximal lifetime number of 3 previous suicide attempts, including the most recent);
* 50 Affective controls, i.e. currently depressed patients without any lifetime history of suicide attempt;
* 50 Healthy controls (age- and gender-matched to patients' groups) with no lifetime history of psychiatric disorders.

The protocol includes two visits for patients (suicide attempters and affective controls) and only one visit (inclusion) for healthy controls.

The first visit is the inclusion visit (Day 0-Day 8). Day 0 is the date of the last suicide attempt for the suicide attempters group and the date of signature of the consent for the affective control and healthy control groups. All the visit exams will be performed within 8 days after Day 0.

The second visit takes place one month +/- one week after inclusion. At each visit, a clinical assessment will be performed to characterise psychopathology and suicidal characteristics. Blood samples will be obtained in order to measure inflammatory markers. An MRI will be performed on order to study white matter microstructure and brain functional connectivity networks.

ELIGIBILITY:
Common inclusion criteria:

* Aged between 18 and 55 years old,
* Affiliated to a French National Social Security System
* Able to understand the nature, purpose and methodology of the study
* Able to give written informed consent

Specific inclusion criteria

Suicide attempters:

* Subject with a main psychiatric diagnosis of current major depressive episode according to DSM-5 criteria (the existence of psychiatric comorbidities is not a non-inclusion criterion)
* Subject with a recent history of proven suicide attempt (within the 8 days before inclusion)
* Subject with a history of maximum 2 previous lifetime proven SA

Affective controls:

* Subject with a main psychiatric diagnosis of current major depressive episode according to DSM-5 criteria (the existence of psychiatric comorbidities is not a non-inclusion criterion),
* Subject without any lifetime history suicidal behavior (proven, interrupted or aborted)

Healthy controls:

- Subject who have no current or past personal history of psychiatric disorders according to DSM5 criteria.

Non inclusion criteria

* History of psychotic disorders
* Diagnostic of illicit substance / alcohol use disorder within the last 6 months
* Current inflammation-related symptoms including fever and infectious or inflammatory disease
* Severe symptomatic or unstable medical condition (e.g., unstable endocrine or cardiovascular disease)
* Medical disorders affecting CNS function (e.g., history of severe head trauma, epilepsy, tumor)
* Current use of specific medications known to affect the immune system, such as corticosteroids, non-steroid anti-inflammatory drugs, aspirin and statins
* Contraindication to MRI or impossibility to assess, or doubt about a contraindication to the MRI: metallic artificial heart valve, pacemaker, cerebrovascular clips ferromagnetic materials, metallic foreign body that can be mobilized, in particular cerebral or intraocular, prosthesis ferromagnetic, impossibility of absolute immobility in supine position, claustrophobia.
* Vaccination in the last month
* Law protected or deprived of liberty subject
* Pregnant and breastfeeding women
* BMI > 30 kg/m2
* Having reached 6000€ annual compensation for participating to clinical trials
* Being in exclusion period for another study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Level of blood S100B assayed in the 3 groups, a marker of cerebral and vascular lesions. | At inclusion
Level of blood S100B assayed in the 3 groups, a marker of cerebral and vascular lesions. | At 1 month follow-up

SECONDARY OUTCOMES:
Cytokines' concentration by multiplex ELISA (pg/ml) | At inclusion
  C-C motif chemokine ligand (CCL)2, CCL3, CCL4, CCL11, CCL13, CCL17, CCL20, CCL22, CCL26, C-X-C motif chemokine ligand (CXCL)10, Interleukin (IL)-1α, IL 1ß, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12/IL-23 p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IL- 27, IL-31, interferon (IFN)-γ, Tumor Necrosis Factor ðTNFÞ α, TNF ß and Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF)
Cytokines' concentration by multiplex ELISA (pg/ml) | At 1 month follow-up
  C-C motif chemokine ligand (CCL)2, CCL3, CCL4, CCL11, CCL13, CCL17, CCL20, CCL22, CCL26, C-X-C motif chemokine ligand (CXCL)10, Interleukin (IL)-1α, IL 1ß, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12/IL-23 p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IL- 27, IL-31, interferon (IFN)-γ, Tumor Necrosis Factor ðTNFÞ α, TNF ß and Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF)
Specific proteins measurement (pg/ml) | At inclusion
  Specific proteins measurement (i.e. GFAP, NFL, UHC-L1, sGPR56, S100B, MBP and related proteins) using digital or classical ELISA or western blot
Specific proteins measurement (pg/ml) | At 1 month follow-up
  Specific proteins measurement (i.e. GFAP, NFL, UHC-L1, sGPR56, S100B, MBP and related proteins) using digital or classical ELISA or western blot
FACS analysis on fresh blood | At inclusion
  Determination of the number of white cells
FACS analysis on fresh blood | At 1 month follow-up
  Determination of the number of white cells
FACS analysis on fresh blood | At inclusion
  Description of the phenotype of white cells
FACS analysis on fresh blood | At 1 month follow-up
  Description of the phenotype of white cells
FACS analysis on fresh blood | At inclusion
  Percentage of cellular inflammatory marker
FACS analysis on fresh blood | At 1 month follow-up
  Percentage of cellular inflammatory marker
Extraction of small and long RNA | At inclusion
  Use of RNA-seq, RT-qPCR and digital PCR to quantify RNA
Extraction of small and long RNA | At 1 month follow-up
  Use of RNA-seq, RT-qPCR and digital PCR to quantify RNA
Test of the capacity of leukocytes isolated from patients to provoke vascular inflammation and BBB permeabilization | At inclusion
  These experiments will be performed using an in vitro model of vascular cell co-culture. The reactivity of leukocytes to pro-inflammatory challenges and cytokines will be tested.
Test of the capacity of leukocytes isolated from patients to provoke vascular inflammation and BBB permeabilization | At 1 month follow-up
  These experiments will be performed using an in vitro model of vascular cell co-culture. The reactivity of leukocytes to pro-inflammatory challenges and cytokines will be tested.
White matter microstructure analysis | At inclusion
  The ihMT (ihMTR) and MT (MTR) ratios will be performed in the apparently normal white and gray matter regions from regional white matter and gray matter atlases
White matter microstructure analysis | At 1 month follow-up
  The ihMT (ihMTR) and MT (MTR) ratios will be performed in the apparently normal white and gray matter regions from regional white matter and gray matter atlases
White matter microstructure analysis | At inclusion
  Value of the fraction of anisotropy (FA) along the skeleton of the Tract-based spatial statistics TBSS
White matter microstructure analysis | At 1 month follow-up
  Value of the fraction of anisotropy (FA) along the skeleton of the Tract-based spatial statistics TBSS
White matter microstructure analysis | At inclusion
  Extraction by anatomical region of FA, mean, axial and radial diffusivity [FSL software)
White matter microstructure analysis | At 1 month follow-up
  Extraction by anatomical region of FA, mean, axial and radial diffusivity [FSL software)
White matter microstructure analysis | At inclusion
  Value of diffusion of blood water D* (pseudocoefficient =perfusive composante) from different region based on regional atlases
White matter microstructure analysis | At 1 month follow-up
  Value of diffusion of blood water D* (pseudocoefficient =perfusive composante) from different region based on regional atlases
White matter microstructure analysis | At inclusion
  Value of diffusion of the tissue (ADC) from different region based on regional atlases
White matter microstructure analysis | At 1 month follow-up
  Value of diffusion of the tissue (ADC) from different region based on regional atlases
White matter microstructure analysis | At inclusion
  Value of fraction of perfusion fD* ( incoherent blood signal divided by total incoherent signal) from different region based on regional atlases
White matter microstructure analysis | At 1 month follow-up
  Value of fraction of perfusion fD* ( incoherent blood signal divided by total incoherent signal) from different region based on regional atlases
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At inclusion
  Regional homogeneity
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At 1 month follow-up
  Regional homogeneity
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At inclusion
  Amplitude of low frequency fluctuations
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At 1 month follow-up
  Amplitude of low frequency fluctuations
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At inclusion
  Functional homotopy
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At 1 month follow-up
  Functional homotopy
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At inclusion
  Graph theory metrics
Brain functional connectivity networks analysis : extraction of resting state functional connectivity metrics from functional atlas or by voxel | At 1 month follow-up
  Graph theory metrics
Cerebral morphometric extraction (3DT1): automatic segmentation | At inclusion
  Evaluation of the volume from cerebral anatomical atlas
Cerebral morphometric extraction (3DT1): automatic segmentation | At 1 month follow-up
  Evaluation of the volume from cerebral anatomical atlas
Cerebral morphometric extraction (3DT1): automatic segmentation | At inclusion
  Evaluation of the surface from cerebral anatomical atlas
Cerebral morphometric extraction (3DT1): automatic segmentation | At 1 month follow-up
  Evaluation of the surface from cerebral anatomical atlas
Cerebral morphometric extraction (3DT1): automatic segmentation | At inclusion
  Evaluation of the cortical thickness from cerebral anatomical atlas
Cerebral morphometric extraction (3DT1): automatic segmentation | At 1 month follow-up
  Evaluation of the cortical thickness from cerebral anatomical atlas
Cerebral blood analysis | At inclusion
  Extraction of blood flow values from 3D PCASL acquisition from vascular atlas
Cerebral blood analysis | At 1 month follow-up
  Extraction of blood flow values from 3D PCASL acquisition from vascular atlas

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Montpellier, France